CLINICAL TRIAL: NCT04994951
Title: Pilot Study of Traditional Chinese Medicine (Qing-Re-Liang-Xue Decoction) as Complementary Medicine for Psoriasis Vulgaris of Blood-heat Syndrome.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Pujiang Hospital of Traditional Chinese Medicine (Unknown); Yongkang Hospital of Traditional Chinese Medicine (Unknown); Ningbo Hospital of Traditional Chinese Medicine (Unknown); Wenzhou Hospital of Integrated Traditional Chinese and Western Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KLJ-001-02
Record Dates: First submitted 2021-07-14; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qing-Re-Liang-Xue Decoction. (Experimental): One dose of granules is mixed, poured into 500ml of boiling water, and taken twice in the morning and afternoon. Women stop taking Chinese medicine during the first 3 days of menstruation. Triamcinolone Acetonide Acetate and Urea Cream,10g/tube and Calcipotriol Ointment,10g/tube are used alternately. The period of treatment will be 10 weeks.
  Interventions: Drug: Qing-Re-Liang-Xue Decoction.
- control group (Active Comparator): Topical steroids. Triamcinolone Acetonide Acetate and Urea Cream,10g/tube and Calcipotriol Ointment,10g/tube are used alternately. The period of treatment will be 10 weeks.
  Interventions: Drug: Triamcinolone Acetonide Acetate and Urea Cream.

INTERVENTIONS:
Drug: Triamcinolone Acetonide Acetate and Urea Cream. — 10g/tube and CalcipotriolOintment,10g/tube are used alternately.
  Arms: control group
Drug: Qing-Re-Liang-Xue Decoction. — One dose of granules is mixed, poured into 500ml of boiling water, and taken twice in the morning and afternoon. Women stop taking Chinese medicine during the first 3 days of menstruation.The period of treatment will be 10 weeks.
  Arms: Qing-Re-Liang-Xue Decoction.

SUMMARY:
Psoriasis is a non-contagious erythematous scaly skin disease characterized by epidermal proliferation and inflammation. The etiology is related to heredity, infection, allergies, metabolic disorders and autoimmunity. The incidence of psoriasis in the survey was about 1.2‰ in 1984 in China, and 2.6% in the United States. In recent years, the incidence of psoriasis has been on the increase trend, mostly in the young to middle age adults, and it can last a lifetime. The characteristic of the disease is that it usually spreads all over the body, or gradually aggravates, or is fixed and difficult to subside,or the disease course is long, lingering and difficult to heal, and it brings great harm to the patient's body and mind. At present, there is no effective treatment for psoriasis. Although western medicine has good short-term curative effects, prolonged use is not advocated because of adverse side effects and poor long-term effects. Besides, it is easy to relapse and aggravate after stopping the medicine. Psoriasis belongs to the category of "baibi" in Chinese medicine. Doctors of the past dynasties mostly treated it from blood heat, blood stasis, and blood deficiency syndrome. Researcher Zhu Renkang believes that "blood with heat" is the main cause of psoriasis and famous TCM dermatologists such as Zhang Zhili, Gu Bohua, Xu Yihou and others all regard "blood-heat syndrome" as the basic pathogenesis of psoriasis. We used Qingre Liangxue Recipe Granules to observe the treatment of 31 patients with blood-heat type psoriasis vulgaris, and found that the PASI index of the patients after treatment was significantly lower than before treatment (P <0.01), and the serum VEGF level was significantly decreased (P < 0.01), the correlation analysis between the two showed a significant correlation. This study aims to further evaluate the efficacy and safety of Qing-Re-Liang-Xue Decoction in comparison with commonly used glucocorticoids and calcipotriol ointment in patients with blood-heat type psoriasis vulgaris.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-label, controlled pilot study of Traditional Chinese medicine (Qing-Re-Liang-Xue Decoction) as a complementary therapy to treat psoriasis vulgaris of blood-heat syndrome during a 10-week period. We estimate to enroll 200 subjects (treatment group(N=100); controlled group(N=100)).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years;
* Had a diagnosis of psoriasis vulgaris for ≥6 months;
* TCM syndrome evaluation belongs to blood-heat type patients: it is more common in the advanced stage of psoriasis. Symptoms: skin lesions develop faster, skin lesions are bright red, blood loss is obvious, scales are dry and thick, itching is severe; upset, and thirsty, dry stool; red-purple tongue, yellow fur, string or slippery or rapid pulse;
* Patients without serious primary diseases, such as cardiovascular, cerebrovascular, liver, kidney and hematopoietic system or mental illnesses;
* Those who are willing to cooperate and can persist in the treatment without interruption;
* During the treatment period, those who have not taken or used other psoriasis drugs externally.

Exclusion Criteria:

* Patients with serious primary diseases, such as cardiovascular, cerebrovascular, liver, kidney and hematopoietic system or mental illnesses;
* History of immunosuppressant medication in the past three months;
* Those who use other drugs during treatment or stop treatment on their own and have incomplete observation data;
* Pregnancy or risk of pregnancy, and/or lactation;
* Aged ≤18 or ≥65 years old;
* Patients with other types of psoriasis, such as articular, pustular, and erythroderma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
participants achieving either a major clinical response or partial clinical response defind by Psoriasis Area Severity Index (PASI) over the 10 weeks treatment period. | 10 weeks
  Psoriasis Area Severity Index (PASI) is usually used to measure the clinical activity diseases of psoriasis.

SECONDARY OUTCOMES:
Changes in skin lesions are assessed by dermoscope. | 10 weeks.
  Image data of skin lesions, capillaries in the nail bed, capillaries near the wing of the nose, etc will be analyzed by the Image-Pro Plus software(Version 6.0，Media Cybernetics) to figure out the inner diameter of the blood vessel wall thickness ratio, Wall cavity cross-sectional area ratio and density.
Evaluation of curative effect of Traditional Chinese medicine is assessed by patient reported outcome(PRO) and clinician reported outcomes(CRO). | 10 weeks.
  Healed: TCM syndromes and skin lesions disappeared, only pigmentation spots or depigmentation spots remained, and no new skin rashes. The TCM syndrome score is reduced by more than 90%; markedly effective: TCM syndromes and skin lesions have basically disappeared or only a few intractable small pieces remain, and the skin lesions are still slightly infiltrated. TCM syndrome scores are reduced by 60-89%; effective: TCM syndromes are significantly reduced, and skin lesions have subsided by more than 30%. TCM syndrome scores are reduced by 30-56%; ineffective: after 3 courses of treatment, the skin lesions still have no progress or the skin lesions have subsided by less than 30%. The reduction of TCM syndrome points is less than 30%.
Compliance evaluation is assessed by Counting Days of Treatment. | 10 weeks.
  Compliance=The number of days the subject has received treatment/The number of days the subject should receive treatment*100%

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No